CLINICAL TRIAL: NCT05075460
Title: A Prospective, Multicenter, Phase III, Non-randomized Study of Tucidinostat, Azacitidine Combined With CHOP Versus CHOP in Patients With Untreated Peripheral T-cell Lymphoma
Brief Title: Tucidinostat, Azacitidine Combined With CHOP Versus CHOP in Patients With Untreated Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhang, MD, Deputy Chief Physician, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-010
Record Dates: First submitted 2021-09-22; First posted 2021-10-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: T-cell Lymphoma
Keywords: Tucidinostat; Azacitidine; CHOP
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tucidinostat, Azacitidine combined with CHOP (Experimental): Tucidinostat, Azacitidine combined with CHOP
  Interventions: Drug: Tucidinostat, Azacitidine combined with CHOP
- CHOP (Active Comparator): CHOP
  Interventions: Drug: Tucidinostat, Azacitidine combined with CHOP

INTERVENTIONS:
Drug: Tucidinostat, Azacitidine combined with CHOP — Azacitidine: 200 mg D1200 mg D2100 mg D3 subcutaneous injection Tucidinostat: 20mg / time, D1, 4, 8, 11; Take medicine with 200ml warm boiled water 30 minutes after breakfast.
  CHOP chemotherapy:
  * Cyclophosphamide (CTX) 750mg / m2 intravenous infusion, day 1;
  * Epirubicin (EPI) 70mg / m2 intravenous infusion, day 1;
  * Vinoresin (VDS) 4mg intravenous infusion, day 1;
  * Prednisone 100mg orally, day 1-5. Every 21 days is a course of treatment

SUMMARY:
This is a prospective, multicenter, phase III study of Tucidinostat, Azacitidine combined with CHOP versus CHOP in patients with untreated peripheral T-cell lymphoma

DETAILED DESCRIPTION:
Tucidinostat, a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. Azacytidine is a hypomethylating agent. The aim of this study is to compare the efficacy and safety of azacytidine, tucidinostat combined with CHOP regimen and classical CHOP regimen in the treatment of primary PTCL

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral T-cell lymphoma confirmed by primary pathology;
* Age 18-70 years;
* ECOG performance status ≤ 2;
* Adequate bone marrow hematopoietic function: WBC > 3.5 × 10*9/L，ANC>1.5 × 10*9/L，HGB>90g/L，PLT>80 × 10*9/L;
* Adequate organ function: cardiac function grade 0-2 (NYHA); SpO2 > 88% (natural condition); ALT<3UNL，TBil<2ULN; SCr>60ml/min/m2;
* Patients have signed the Informed Consent Form

Exclusion Criteria:

* ALK positive anaplastic T-cell lymphoma;
* NK / T cell lymphoma, nasal type;
* Uncontrolled active infection;
* Acute myocardial infarction or unstable angina pectoris within 6 months; uncontrolled hypertension, symptomatic arrhythmia, etc;
* Subjects who are known or suspected to be unable to comply with the study protocol;
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 course of treatment (each cycle is 21 days)
  the total proportion of patients with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
2-year progression-free survival（PFS） | 2 years
  Time from treatment until disease progression or death
2-year overall survival（OS） | 2 years
  Time from treatment until death from any cause
Incidence and severity of adverse events, serious adverse events and other safety parameters | 2 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, Study Chair — Department of Hematology, Peking University First Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China